CLINICAL TRIAL: NCT01010412
Title: Ultrasound Visualization v. Electrical Nerve Stimulation for the Safety and Effectiveness of Interscalene/Axillary Nerve Block in Upper Extremity Surgery: A Randomized Trial
Brief Title: Ultrasound Visualization Versus Electrical Nerve Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allentown Anesthesia Associates (Other)
Collaborators: SonoSite, Inc. (Industry)
Responsible Party: Principal Investigator, Nanette Schwann, M.D., MD, Allentown Anesthesia Associates
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UVVENS
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Trauma to the Arm, Shoulder, Elbow, Forearm, or Hand
Keywords: Ultrasound; Nerve blocks; Upper extremity
MeSH Terms: interventions — Ultrasonography; Needles

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Ultrasound guided nerve localization through direct visualization of the nerves and surrounding structures.
  Interventions: Device: Ultrasound (Sonosite Titan T-shaped ultrasound probe)
- Nerve Stimulation (Active Comparator): Standard of Care
  Interventions: Device: Electrical Nerve Stimulation (Stimuplex (B Braun) needle)

INTERVENTIONS:
Device: Ultrasound (Sonosite Titan T-shaped ultrasound probe) — Ultrasonography will allow direct visualization of nerves. As local anesthetic is injected, it can be seen surrounding the nerve.
  Other Names: Sonosite Titan T-shaped ultrasound probe
  Arms: Ultrasound
Device: Electrical Nerve Stimulation (Stimuplex (B Braun) needle)
  Arms: Nerve Stimulation

SUMMARY:
Hypothesis and Specific Aims:

The investigators hypothesize that ultrasound (US) visualization is as effective as nerve stimulation (NS) for identification of peripheral nervous structures and may be associated with less trauma and patient discomfort. Specifically, the investigators believe that equivalent rates of surgical anesthesia are achievable with non-invasive ultrasonic needle guidance in comparison to needle guidance by intensity of motor fiber response to intermittent electrical nerve stimulation. Specifically, the number of needle sticks to identify the brachial plexus and total time to plexus sheath injection may be reduced while achieving similar efficacy rates. The investigators hypothesize that similar composite safety and efficacy endpoints but improved patient satisfaction and acceptance will favor US over NS guidance of nerve blocks indicated for surgery on the extremity surgery. However, the investigators believe that an economic assessment based upon capital hardware investment, operating room utilization, total block time, and pay for performance patient satisfaction metrics require examination prior to assimilation of new technology into clinical practice.

DETAILED DESCRIPTION:
This is a prospective randomized study of 450 consecutive patients presenting for upper extremity surgery scheduled to receive NB without general anesthesia for their surgical procedure. Patients will be randomized to receive one of two nerve localization techniques in a 1:1 randomization ratio. Primary intraoperative providers of supplemental sedative, additional local anesthetic infiltration or analgesia, general anesthesia and assessors of VAS or PCI will be blinded to the technique.

Patients over 18 years of age presenting for elective upper extremity surgery planned in the supine position under isolated interscalene or axillary nerve block will be screened. Up to 450 patients undergoing unilateral upper extremity procedures at Lehigh Valley Hospital will be enrolled.

STUDY PROCEDURES Screening:

All patients meeting inclusion criteria and not meeting exclusion criteria will be eligible to be enrolled. All subjects who have preadmission testing will be recruited prior to their surgical procedure with initial contact made before the day of their scheduled surgery. For patients who do not have preadmission testing scheduled and are found to be eligible for the study on the day of surgery, those patients will be consented for the study the morning of their procedure by the study anesthesiologist. Only patients who are able to understand English and who are able to legally give written informed consent will be recruited to the study. Following signed informed consent (IRB approved) and permission of their surgeon and anesthesiologist and prior to the start of anesthesia, vital signs, standard lab tests, patient history and physical examination will be reviewed.

Day of Procedure:

For the NS group, interscalene/axillary block will be performed in the standard method using a nerve stimulator attached to a four centimeter Stimuplex (B Braun) needle. Following application of routine monitors, supplemental oxygen via facemask, and intravenous sedation, the skin overlying the brachial plexus will be anesthetized. The Stimuplex needle will then be inserted and guided into a position in close proximity to the brachial plexus using an endpoint of muscle twitches involving the hand at a stimulus intensity of less than 0.5 milliamps to the satisfaction of the operator. Forty (40) milliliters of 0.5 percent Bupivicaine with 1.5% Mepivicaine with 1:200,00 of epinephrine will be injected incrementally with intermittent aspiration. This block is chosen for the study because of its widespread use for a variety of shoulder procedures and for its low incidence of complications. The quoted success rate in the literature for interscalene block ranges from 70 to 95 percent.

For the US group interscalene block will be performed in a method using ultrasound guided needle insertion. Following application of routine monitors, supplemental oxygen via facemask, and intravenous sedation, the skin overlying the brachial plexus will be anesthetized. A sterile cover will be used for the ultrasound probe. Using this probe, the anesthesiologist can visualize the nerve and will maneuver the tip of the needle into the nerve guided by the of ultrasound probe. Forty (40) milliliters of 0.5% Bupivicaine with 1.5% Mepivicaine with 1:200,00 of Epinephrine will be injected incrementally with intermittent aspiration. This block is chosen for the study because of its widespread use for a variety of shoulder procedures and for its low incidence of complications. The quoted success rate in the literature for interscalene block ranges for 70 to 95 percent.

The brachial plexus will be visualized at the level of the roots of the plexus at this level. Presence or absence of local anesthetic around the nerves will be recorded using a Sonosite Titan T-shaped ultrasound probe placed on the patient's skin. Still images of the brachial plexus and the local anesthetic will be captured for each patient. Patient identifiers will be on the images, however the images are placed on the patient's medical record.

Assessment of block success:

The success of the block will be assessed by examining motor strength in the anesthetized extremity and degree of anesthesia at 30 minutes after injection. Strength in the distribution of the musculocutaneous, median, radial, and ulnar nerves will be assessed. Pinprick and cold sensation will be assessed in the same distributions. A successful block will be one with a lack of sensation to cold and pinprick in the above distributions as well as strength less than three out of five on the standard scale of strength testing in all of the above distributions. Ultimately, block success (yes/no) will be determined by pain free surgery not requiring general anesthesia. The patient comfort index and post op assessments will be carried out as above.

Completion of the Study:

The study will be complete at PACU discharge after the patient returns his/her assessment of PCI and pain and nausea data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 years of age at the time of screening
* ASA Class I - IV, undergoing unilateral elective surgical procedure involving the shoulder, arm, elbow, forearm, or hand
* Planned interscalene block

Exclusion Criteria:

* Peripheral neuropathy
* Coagulopathy
* Anticoagulant treatment that would preclude regional anesthesia
* Local anesthetic allergy
* Infection at the site of injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Successful Block: defined by avoidance of General Anesthesia (which will be documented in the medical record as such) | 30 minutes after injection

SECONDARY OUTCOMES:
Amount of sedation required for block. (mg of drug) | 30 minutes after injection

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Schwann, M.D., Principal Investigator — Allentown Anesthesia Associates
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States

REFERENCES:
- [Background] Gray AT, Schafhalter-Zoppoth I. Ultrasound guidance for ulnar nerve block in the forearm. Reg Anesth Pain Med. 2003 Jul-Aug;28(4):335-9. doi: 10.1016/s1098-7339(03)00196-2. PMID 12945028